CLINICAL TRIAL: NCT01679431
Title: Metabolic Determinants of the Progression of Aortic Stenosis - PROGRESSA Study
Brief Title: Metabolic Determinants of the Progression of Aortic Stenosis
Acronym: PROGRESSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Philippe Pibarot, Doctor, Laval University
Other Study IDs: MOP-114997
Record Dates: First submitted 2012-08-24; First posted 2012-09-06 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Stenosis; Obesity, Abdominal; Metabolic Syndrome X; Insulin Resistance; Echocardiography, Doppler; Multidetector Computed Tomography; Magnetic Resonance Imaging
MeSH Terms: conditions — Aortic Valve Stenosis; Obesity, Abdominal; Metabolic Syndrome; Insulin Resistance | interventions — Echocardiography, Doppler; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fasting blood sample (serum, lithium-heparin, EDTA) and white cells - Tissue (explanted aortic valves)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with aortic stenosis: Patients have every year: 1) an assessment of cardiometabolic risk profile with measure of body mass index, waist circumference and fasting blood sample and 2) a comprehensive Doppler-echocardiography exam.
  Computed tomography and magnetic resonance imaging are performed every 2 years.
  Interventions: Diagnostic Test: Doppler-echocardiography; Radiation: Computed tomography; Other: Magnetic resonance imaging; Biological: Fasting blood sample

INTERVENTIONS:
Diagnostic Test: Doppler-echocardiography
Radiation: Computed tomography
Other: Magnetic resonance imaging
Biological: Fasting blood sample

SUMMARY:
Calcific aortic stenosis (AS) has become the most common cardiac disease after coronary artery disease and hypertension. Unfortunately no medical therapies have been proven to decrease either the progression of valve stenosis or the resulting adverse effects on myocardial remodeling and function. In light of the studies performed in PROGRESSA, it becomes obvious that: i) AS is a complex and actively regulated process that involves the interaction of several pathways including lipid infiltration and retention, chronic inflammation, osteogenic activation, and active mineralization within the valvular tissues; ii) AS is not a disease strictly limited to the aortic valve but rather a systemic disease that often involves calcification and stiffening of the aorta and impairment of LV function as a consequence of pressure overload. Our findings suggest that the dysmetabolic milieu linked to visceral obesity may accelerate the deterioration of the structure and function not only of the aortic valve but also of the aorta and of the left ventricle. These findings open new avenues of research and provide strong impetus for the elaboration of prospective studies focusing on the "valvulo-metabolic risk" in AS.

The general hypotheses are: The metabolic abnormalities linked to visceral obesity accelerate (1) the progression of valvular calcification and stenosis, aortic calcification and stiffness; (2) the progression of myocardial fibrosis and dysfunction.

The general objectives of the study are to elucidate the mechanisms implicated in the pathogenesis of AS and to identify the metabolic factors that determine the progression of: i) aortic valve calcification and stenosis; ii) myocardial fibrosis and dysfunction; and iii) clinical outcomes.

This study will contribute to identifying the key metabolic determinants of AS progression and will pave the way for the future development of non surgical therapies for this disease. The results of this study would provide strong support to the realization of randomized trial to test the efficacy of lifestyle modification program or new pharmacological treatment aiming at the reduction of visceral fat and associated metabolic abnormalities in the AS population. Furthermore, this study will contribute to the identification of novel blood and imaging biomarkers of faster disease progression, which will help to optimize risk stratification and timing of AVR in the AS population.

DETAILED DESCRIPTION:
The hypotheses are: (1) The metabolic abnormalities linked to visceral obesity increase: i) the progression of aortic valve calcification and stenosis, of aortic calcification and stiffness, and thereby of the global hemodynamic load imposed on the LV; ii) the progression of myocardial hypertrophy, fibrosis, and dysfunction, iii) the loss in bone mineral density, and iv) the occurrence of adverse events in patients with AS. (2) Specifically, insulin resistance, the small, dense LDL and HDL phenotypes, enhanced oxidative stress & inflammatory state, and activation of the RAS act synergistically to: i) promote infiltration, retention, and modification of lipids within the valvular and arterial tissues, ii) enhance the inflammatory and osteoblastic response to oxidized lipids, iii) activate apoptosis of VICs and apoptosis-mediated calcification of the aortic valve and aorta, iv) promote osteoclastic activity and demineralization within the bone tissues (calcification paradox) (Figs. 1&6). These mechanisms predominate in the middle-aged patients, whereas imbalance in nuclear coregulators, alteration of adipokine system, dysregulation of mineral metabolism, and loss calcification inhibitors are the main contributing mechanisms in the elderly (Figs. 1,5,6). The contribution of visceral obesity to disease progression is more important in the patients with mildly or moderately calcified valves than in those with heavily calcified valves. In the latter, further progression of calcification and stenosis is predominantly influenced dysregulation of mineral metabolism. (3) The alteration of the myocardial energetic substrates and of the protein synthesis/degradation balance associated with visceral obesity and insulin resistance amplify the development of myocardial hypertrophy and fibrosis in response to pressure overload and accelerates the progression to myocardial dysfunction (Figs. 7&8). The adverse LV remodelling and fibrosis resulting from the synergistic effects of pressure overload and dysmetabolism predispose to the occurrence of paradoxical low flow AS and cardiac events.

The general objectives of the study are to elucidate the mechanisms implicated in the pathogenesis of AS and to identify the metabolic factors that determine the progression of: i) aortic valve calcification and stenosis; ii) aorta calcification and stiffness, iii) myocardial remodeling, fibrosis and dysfunction; and iv) clinical outcomes in the AS population.

The specific aims of the study are:

1. To obtain and analyze: i) the metabolic profile, ii) the progression of aortic valve, aorta, and coronary artery calcification measured by CT, iii) the hemodynamic progression of valve stenosis by Doppler-echocardiography, iv) the progression of myocardial remodeling, fibrosis, and dysfunction by MRI, v) the change in bone mineral density by DXA, vi) the occurrence of clinical outcomes (AVR or death), and vii) the valvular tissues explanted at the time of AVR in a series of 280 patients with AS.
2. To perform histo-pathologic and genetic/protein expression analyses of valve tissues to document the lipid infiltration /retention/modification and the inflammatory and osteoblastic activities within the metabolic abnormalities, age, valve phenotype, and bone mineral density.
3. To study the relationship between the cardio-metabolic determinants: i) traditional cardiovascular risk factors (hypercholesterolemia, hypertension, smoking), ii) amount of visceral fat and metabolic abnormalities associated with visceral obesity and the outcome variables: i) progression of aortic valve calcification and stenosis, aorta calcification and stiffening, bone mineral loss, and myocardial remodelling, fibrosis and dysfunction, ii) occurrence of adverse outcomes, iii) lipid infiltration/ retention/ modification, inflammatory/osteoblastic activities in the valve
4. To determine if the impact of these cardio-metabolic determinants on disease progression differ according to age, gender, BAV phenotype, and degree of aortic valve calcification at baseline.
5. To examine the relationship between aortic valve/aorta/coronary (i.e. ectopic) calcification and bone mineral density and determine the impact of cardio-metabolic and mineral metabolism factors on this relationship.
6. To examine the respective contribution of aortic valve calcification/stenosis, aorta calcification /stiffness, coronary calcification, bone density, and myocardial fibrosis to the occurrence of clinical outcomes in this AS cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 years
* Presence of aortic stenosis defined as peak aortic jet velocity ≥2.5 m/s

Exclusion Criteria:

* Symptomatic aortic stenosis
* Very severe aortic stenosis defined as an AVA≤0.6 cm2
* Left ventricular ejection fraction < 50%
* More than mild aortic or mitral regurgitation, or mitral stenosis
* Atrial fibrillation or flutter
* Pregnant or lactating women
* Contraindications to gadolinium-enhanced MRI

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort will be selected at primary care clinic
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2005-04; Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Progression of aortic valve stenosis | Patients will be followed every 1 year, up to 5 years
  Annualized progression rate of aortic stenosis hemodynamic severity calculate as the difference between peak aortic jet velocity, transvalvular gradients, and aortic valve area measured at baseline and those measured at the last follow-up divided by the time between the first and last examinations.

SECONDARY OUTCOMES:
Progression of aortic valve calcification | Patients will be followed every 2 years, up to 5 years
  Annualized progression rate of aortic valve calcium
Progression of myocardial fibrosis and dysfunction | PPatients will be followed every 2 years, up to 5 years
  Annualized progression rate of myocardial fibrosis and global longitudinal myocardial strain

OTHER OUTCOMES:
Progression of aortic calcification and stiffness | Patients will be followed every 2 years, up to 5 years
  Annualized progression rate of calcification measured by computed tomography and aortic compliance measured (CT) by cardiac magnetic resonance (CMR) and Doppler-echocardiography
Progression of coronary artery calcification | Patients will be followed every 2 years, up to 5 years
  Annualized progression rate of coronary artery calcification measured by CT
Progression of global hemodynamic load | Patients will be followed every 1 year, up to 5 years
  Annualized progression rate of valvulo-arterial impedance measured by Doppler-echocardiography
Aortic stenosis related events | From date of baseline until the date of first documented aortic stenosis related events (as defined on description box), assessed up to 5 years
  Cardiovascular-related mortality; hospitalization for heart failure; surgical or transcatheter aortic valve replacement motivated by the development of symptoms or LV systolic dysfunction
Ischemic cardiovascular events | From date of baseline until the date of first documented ischemic cardiovascular events (as defined on description box), assessed up to 5 years
  Myocardial infarction; unstable angina; revascularization procedure
All-cause mortality | From date of baseline until the date of death from any cause assessed up to 5 years
  Death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Pibarot, PhD, DVM, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Canada

REFERENCES:
- [Background] Capoulade R, Clavel MA, Dumesnil JG, Chan KL, Teo KK, Tam JW, Cote N, Mathieu P, Despres JP, Pibarot P; ASTRONOMER Investigators. Impact of metabolic syndrome on progression of aortic stenosis: influence of age and statin therapy. J Am Coll Cardiol. 2012 Jul 17;60(3):216-23. doi: 10.1016/j.jacc.2012.03.052. PMID 22789885
- [Background] Cote N, El Husseini D, Pepin A, Bouvet C, Gilbert LA, Audet A, Fournier D, Pibarot P, Moreau P, Mathieu P. Inhibition of ectonucleotidase with ARL67156 prevents the development of calcific aortic valve disease in warfarin-treated rats. Eur J Pharmacol. 2012 Aug 15;689(1-3):139-46. doi: 10.1016/j.ejphar.2012.05.016. Epub 2012 May 31. PMID 22659116
- [Background] Audet A, Cote N, Couture C, Bosse Y, Despres JP, Pibarot P, Mathieu P. Amyloid substance within stenotic aortic valves promotes mineralization. Histopathology. 2012 Oct;61(4):610-9. doi: 10.1111/j.1365-2559.2012.04265.x. PMID 22642224
- [Background] Carter S, Miard S, Roy-Bellavance C, Boivin L, Li Z, Pibarot P, Mathieu P, Picard F. Sirt1 inhibits resistin expression in aortic stenosis. PLoS One. 2012;7(4):e35110. doi: 10.1371/journal.pone.0035110. Epub 2012 Apr 6. PMID 22493735
- [Background] Shetty R, Girerd N, Cote N, Arsenault B, Despres JP, Pibarot P, Mathieu P. Elevated proportion of small, dense low-density lipoprotein particles and lower adiponectin blood levels predict early structural valve degeneration of bioprostheses. Cardiology. 2012;121(1):20-6. doi: 10.1159/000336170. Epub 2012 Feb 25. PMID 22378142
- [Background] Cote N, El Husseini D, Pepin A, Guauque-Olarte S, Ducharme V, Bouchard-Cannon P, Audet A, Fournier D, Gaudreault N, Derbali H, McKee MD, Simard C, Despres JP, Pibarot P, Bosse Y, Mathieu P. ATP acts as a survival signal and prevents the mineralization of aortic valve. J Mol Cell Cardiol. 2012 May;52(5):1191-202. doi: 10.1016/j.yjmcc.2012.02.003. Epub 2012 Feb 16. PMID 22366713
- [Background] Cote N, Couture C, Pibarot P, Despres JP, Mathieu P. Angiotensin receptor blockers are associated with a lower remodelling score of stenotic aortic valves. Eur J Clin Invest. 2011 Nov;41(11):1172-9. doi: 10.1111/j.1365-2362.2011.02522.x. PMID 21988540
- [Background] Gaudreault N, Ducharme V, Lamontagne M, Guauque-Olarte S, Mathieu P, Pibarot P, Bosse Y. Replication of genetic association studies in aortic stenosis in adults. Am J Cardiol. 2011 Nov 1;108(9):1305-10. doi: 10.1016/j.amjcard.2011.06.050. Epub 2011 Aug 18. PMID 21855833
- [Background] Mohty D, Pibarot P, Cote N, Cartier A, Audet A, Despres JP, Mathieu P. Hypoadiponectinemia is associated with valvular inflammation and faster disease progression in patients with aortic stenosis. Cardiology. 2011;118(2):140-6. doi: 10.1159/000327588. Epub 2011 May 19. PMID 21597293
- [Background] Page A, Dumesnil JG, Clavel MA, Chan KL, Teo KK, Tam JW, Mathieu P, Despres JP, Pibarot P; ASTRONOMER Investigators. Metabolic syndrome is associated with more pronounced impairment of left ventricle geometry and function in patients with calcific aortic stenosis: a substudy of the ASTRONOMER (Aortic Stenosis Progression Observation Measuring Effects of Rosuvastatin). J Am Coll Cardiol. 2010 Apr 27;55(17):1867-74. doi: 10.1016/j.jacc.2009.11.083. PMID 20413039
- [Background] Derbali H, Bosse Y, Cote N, Pibarot P, Audet A, Pepin A, Arsenault B, Couture C, Despres JP, Mathieu P. Increased biglycan in aortic valve stenosis leads to the overexpression of phospholipid transfer protein via Toll-like receptor 2. Am J Pathol. 2010 Jun;176(6):2638-45. doi: 10.2353/ajpath.2010.090541. Epub 2010 Apr 9. PMID 20382708
- [Background] Bosse Y, Miqdad A, Fournier D, Pepin A, Pibarot P, Mathieu P. Refining molecular pathways leading to calcific aortic valve stenosis by studying gene expression profile of normal and calcified stenotic human aortic valves. Circ Cardiovasc Genet. 2009 Oct;2(5):489-98. doi: 10.1161/CIRCGENETICS.108.820795. Epub 2009 Jul 8. PMID 20031625
- [Background] Cote N, Pibarot P, Pepin A, Fournier D, Audet A, Arsenault B, Couture C, Poirier P, Despres JP, Mathieu P. Oxidized low-density lipoprotein, angiotensin II and increased waist cirumference are associated with valve inflammation in prehypertensive patients with aortic stenosis. Int J Cardiol. 2010 Dec 3;145(3):444-9. doi: 10.1016/j.ijcard.2009.05.054. Epub 2009 Jun 13. PMID 19525020
- [Background] Mohty D, Pibarot P, Despres JP, Cartier A, Arsenault B, Picard F, Mathieu P. Age-related differences in the pathogenesis of calcific aortic stenosis: the potential role of resistin. Int J Cardiol. 2010 Jul 9;142(2):126-32. doi: 10.1016/j.ijcard.2008.12.068. Epub 2009 Jan 21. PMID 19162347
- [Background] Mathieu P, Despres JP, Pibarot P. The 'valvulo-metabolic' risk in calcific aortic valve disease. Can J Cardiol. 2007 Oct;23 Suppl B(Suppl B):32B-39B. doi: 10.1016/s0828-282x(07)71008-5. PMID 17932585
- [Background] Mohty D, Pibarot P, Despres JP, Cote C, Arsenault B, Cartier A, Cosnay P, Couture C, Mathieu P. Association between plasma LDL particle size, valvular accumulation of oxidized LDL, and inflammation in patients with aortic stenosis. Arterioscler Thromb Vasc Biol. 2008 Jan;28(1):187-93. doi: 10.1161/ATVBAHA.107.154989. Epub 2007 Nov 1. PMID 17975118
- [Background] Cote C, Pibarot P, Despres JP, Mohty D, Cartier A, Arsenault BJ, Couture C, Mathieu P. Association between circulating oxidised low-density lipoprotein and fibrocalcific remodelling of the aortic valve in aortic stenosis. Heart. 2008 Sep;94(9):1175-80. doi: 10.1136/hrt.2007.125740. Epub 2007 Oct 11. PMID 17932090
- [Background] Pibarot P, Dumesnil JG, Mathieu P. [New insight into the treatment of aortic stenosis]. Med Sci (Paris). 2007 Jan;23(1):81-7. doi: 10.1051/medsci/200723181. French. PMID 17212936
- [Background] Briand M, Lemieux I, Dumesnil JG, Mathieu P, Cartier A, Despres JP, Arsenault M, Couet J, Pibarot P. Metabolic syndrome negatively influences disease progression and prognosis in aortic stenosis. J Am Coll Cardiol. 2006 Jun 6;47(11):2229-36. doi: 10.1016/j.jacc.2005.12.073. Epub 2006 May 15. PMID 16750688
- [Background] Charest A, Pepin A, Shetty R, Cote C, Voisine P, Dagenais F, Pibarot P, Mathieu P. Distribution of SPARC during neovascularisation of degenerative aortic stenosis. Heart. 2006 Dec;92(12):1844-9. doi: 10.1136/hrt.2005.086595. Epub 2006 May 18. PMID 16709694
- [Background] Shetty R, Pepin A, Charest A, Perron J, Doyle D, Voisine P, Dagenais F, Pibarot P, Mathieu P. Expression of bone-regulatory proteins in human valve allografts. Heart. 2006 Sep;92(9):1303-8. doi: 10.1136/hrt.2005.075903. Epub 2006 Jan 31. PMID 16449517
- [Background] Briand M, Dumesnil JG, Kadem L, Tongue AG, Rieu R, Garcia D, Pibarot P. Reduced systemic arterial compliance impacts significantly on left ventricular afterload and function in aortic stenosis: implications for diagnosis and treatment. J Am Coll Cardiol. 2005 Jul 19;46(2):291-8. doi: 10.1016/j.jacc.2004.10.081. PMID 16022957
- [Background] Tastet L, Capoulade R, Shen M, Clavel MA, Cote N, Mathieu P, Arsenault M, Bedard E, Tremblay A, Samson M, Bosse Y, Dumesnil JG, Arsenault BJ, Beaudoin J, Bernier M, Despres JP, Pibarot P. ApoB/ApoA-I Ratio is Associated With Faster Hemodynamic Progression of Aortic Stenosis: Results From the PROGRESSA (Metabolic Determinants of the Progression of Aortic Stenosis) Study. J Am Heart Assoc. 2018 Feb 10;7(4):e007980. doi: 10.1161/JAHA.117.007980. PMID 29440006
- [Background] Capoulade R, Larose E, Mathieu P, Clavel MA, Dahou A, Arsenault M, Bedard E, Larue-Grondin S, Le Ven F, Dumesnil JG, Despres JP, Pibarot P. Visceral adiposity and left ventricular mass and function in patients with aortic stenosis: the PROGRESSA study. Can J Cardiol. 2014 Sep;30(9):1080-7. doi: 10.1016/j.cjca.2014.02.007. Epub 2014 Feb 19. PMID 24975192
- [Background] Capoulade R, Mahmut A, Tastet L, Arsenault M, Bedard E, Dumesnil JG, Despres JP, Larose E, Arsenault BJ, Bosse Y, Mathieu P, Pibarot P. Impact of plasma Lp-PLA2 activity on the progression of aortic stenosis: the PROGRESSA study. JACC Cardiovasc Imaging. 2015 Jan;8(1):26-33. doi: 10.1016/j.jcmg.2014.09.016. Epub 2014 Nov 1. PMID 25499129
- [Background] Carter S, Capoulade R, Arsenault M, Bedard E, Dumesnil JG, Mathieu P, Pibarot P, Picard F. Relationship Between Insulin-Like Growth Factor Binding Protein-2 and Left Ventricular Stroke Volume in Patients With Aortic Stenosis. Can J Cardiol. 2015 Dec;31(12):1447-54. doi: 10.1016/j.cjca.2015.04.024. Epub 2015 Apr 30. PMID 26243351
- [Background] Tastet L, Capoulade R, Clavel MA, Larose E, Shen M, Dahou A, Arsenault M, Mathieu P, Bedard E, Dumesnil JG, Tremblay A, Bosse Y, Despres JP, Pibarot P. Systolic hypertension and progression of aortic valve calcification in patients with aortic stenosis: results from the PROGRESSA study. Eur Heart J Cardiovasc Imaging. 2017 Jan;18(1):70-78. doi: 10.1093/ehjci/jew013. Epub 2016 Feb 18. PMID 26896413
- [Background] Shen M, Tastet L, Capoulade R, Larose E, Bedard E, Arsenault M, Chetaille P, Dumesnil JG, Mathieu P, Clavel MA, Pibarot P. Effect of age and aortic valve anatomy on calcification and haemodynamic severity of aortic stenosis. Heart. 2017 Jan 1;103(1):32-39. doi: 10.1136/heartjnl-2016-309665. Epub 2016 Aug 8. PMID 27504001
- [Background] Cote N, Mahmut A, Bosse Y, Couture C, Page S, Trahan S, Boulanger MC, Fournier D, Pibarot P, Mathieu P. Inflammation is associated with the remodeling of calcific aortic valve disease. Inflammation. 2013 Jun;36(3):573-81. doi: 10.1007/s10753-012-9579-6. PMID 23225202
- [Background] El Husseini D, Boulanger MC, Fournier D, Mahmut A, Bosse Y, Pibarot P, Mathieu P. High expression of the Pi-transporter SLC20A1/Pit1 in calcific aortic valve disease promotes mineralization through regulation of Akt-1. PLoS One. 2013;8(1):e53393. doi: 10.1371/journal.pone.0053393. Epub 2013 Jan 4. PMID 23308213
- [Background] Mahmut A, Boulanger MC, Fournier D, Couture C, Trahan S, Page S, Arsenault B, Despres JP, Pibarot P, Mathieu P. Lipoprotein lipase in aortic valve stenosis is associated with lipid retention and remodelling. Eur J Clin Invest. 2013 Jun;43(6):570-8. doi: 10.1111/eci.12081. Epub 2013 Apr 1. PMID 23550604
- [Background] Ducharme V, Guauque-Olarte S, Gaudreault N, Pibarot P, Mathieu P, Bosse Y. NOTCH1 genetic variants in patients with tricuspid calcific aortic valve stenosis. J Heart Valve Dis. 2013 Mar;22(2):142-9. PMID 23798201
- [Background] Cote N, Mahmut A, Fournier D, Boulanger MC, Couture C, Despres JP, Trahan S, Bosse Y, Page S, Pibarot P, Mathieu P. Angiotensin receptor blockers are associated with reduced fibrosis and interleukin-6 expression in calcific aortic valve disease. Pathobiology. 2014;81(1):15-24. doi: 10.1159/000350896. Epub 2013 Aug 21. PMID 23969418
- [Background] Garcia J, Capoulade R, Le Ven F, Gaillard E, Kadem L, Pibarot P, Larose E. Discrepancies between cardiovascular magnetic resonance and Doppler echocardiography in the measurement of transvalvular gradient in aortic stenosis: the effect of flow vorticity. J Cardiovasc Magn Reson. 2013 Sep 20;15(1):84. doi: 10.1186/1532-429X-15-84. PMID 24053194
- [Background] Capoulade R, Clavel MA, Mathieu P, Cote N, Dumesnil JG, Arsenault M, Bedard E, Pibarot P. Impact of hypertension and renin-angiotensin system inhibitors in aortic stenosis. Eur J Clin Invest. 2013 Dec;43(12):1262-72. doi: 10.1111/eci.12169. Epub 2013 Oct 7. PMID 24117162
- [Background] Mahmut A, Boulanger MC, El Husseini D, Fournier D, Bouchareb R, Despres JP, Pibarot P, Bosse Y, Mathieu P. Elevated expression of lipoprotein-associated phospholipase A2 in calcific aortic valve disease: implications for valve mineralization. J Am Coll Cardiol. 2014 Feb 11;63(5):460-9. doi: 10.1016/j.jacc.2013.05.105. Epub 2013 Oct 23. PMID 24161325
- [Background] Mahmut A, Mahjoub H, Boulanger MC, Fournier D, Despres JP, Pibarot P, Mathieu P. Lp-PLA2 is associated with structural valve degeneration of bioprostheses. Eur J Clin Invest. 2014 Feb;44(2):136-45. doi: 10.1111/eci.12199. Epub 2013 Nov 28. PMID 24328921
- [Background] Bouchareb R, Boulanger MC, Fournier D, Pibarot P, Messaddeq Y, Mathieu P. Mechanical strain induces the production of spheroid mineralized microparticles in the aortic valve through a RhoA/ROCK-dependent mechanism. J Mol Cell Cardiol. 2014 Feb;67:49-59. doi: 10.1016/j.yjmcc.2013.12.009. Epub 2013 Dec 22. PMID 24368096
- [Background] El Husseini D, Boulanger MC, Mahmut A, Bouchareb R, Laflamme MH, Fournier D, Pibarot P, Bosse Y, Mathieu P. P2Y2 receptor represses IL-6 expression by valve interstitial cells through Akt: implication for calcific aortic valve disease. J Mol Cell Cardiol. 2014 Jul;72:146-56. doi: 10.1016/j.yjmcc.2014.02.014. Epub 2014 Mar 11. PMID 24631773
- [Background] Capoulade R, Magne J, Dulgheru R, Hachicha Z, Dumesnil JG, O'Connor K, Arsenault M, Bergeron S, Pierard LA, Lancellotti P, Pibarot P. Prognostic value of plasma B-type natriuretic peptide levels after exercise in patients with severe asymptomatic aortic stenosis. Heart. 2014 Oct;100(20):1606-12. doi: 10.1136/heartjnl-2014-305729. PMID 24993604
- [Background] Capoulade R, Cote N, Mathieu P, Chan KL, Clavel MA, Dumesnil JG, Teo KK, Tam JW, Fournier D, Despres JP, Pibarot P; ASTRONOMER Investigators. Circulating levels of matrix gla protein and progression of aortic stenosis: a substudy of the Aortic Stenosis Progression Observation: Measuring Effects of rosuvastatin (ASTRONOMER) trial. Can J Cardiol. 2014 Sep;30(9):1088-95. doi: 10.1016/j.cjca.2014.03.025. Epub 2014 Mar 24. PMID 25015689
- [Background] Potus F, Ruffenach G, Dahou A, Thebault C, Breuils-Bonnet S, Tremblay E, Nadeau V, Paradis R, Graydon C, Wong R, Johnson I, Paulin R, Lajoie AC, Perron J, Charbonneau E, Joubert P, Pibarot P, Michelakis ED, Provencher S, Bonnet S. Downregulation of MicroRNA-126 Contributes to the Failing Right Ventricle in Pulmonary Arterial Hypertension. Circulation. 2015 Sep 8;132(10):932-43. doi: 10.1161/CIRCULATIONAHA.115.016382. Epub 2015 Jul 10. PMID 26162916
- [Background] Bouchareb R, Mahmut A, Nsaibia MJ, Boulanger MC, Dahou A, Lepine JL, Laflamme MH, Hadji F, Couture C, Trahan S, Page S, Bosse Y, Pibarot P, Scipione CA, Romagnuolo R, Koschinsky ML, Arsenault BJ, Marette A, Mathieu P. Autotaxin Derived From Lipoprotein(a) and Valve Interstitial Cells Promotes Inflammation and Mineralization of the Aortic Valve. Circulation. 2015 Aug 25;132(8):677-90. doi: 10.1161/CIRCULATIONAHA.115.016757. Epub 2015 Jul 29. PMID 26224810
- [Background] Capoulade R, Chan KL, Yeang C, Mathieu P, Bosse Y, Dumesnil JG, Tam JW, Teo KK, Mahmut A, Yang X, Witztum JL, Arsenault BJ, Despres JP, Pibarot P, Tsimikas S. Oxidized Phospholipids, Lipoprotein(a), and Progression of Calcific Aortic Valve Stenosis. J Am Coll Cardiol. 2015 Sep 15;66(11):1236-1246. doi: 10.1016/j.jacc.2015.07.020. PMID 26361154
- [Background] Guauque-Olarte S, Messika-Zeitoun D, Droit A, Lamontagne M, Tremblay-Marchand J, Lavoie-Charland E, Gaudreault N, Arsenault BJ, Dube MP, Tardif JC, Body SC, Seidman JG, Boileau C, Mathieu P, Pibarot P, Bosse Y. Calcium Signaling Pathway Genes RUNX2 and CACNA1C Are Associated With Calcific Aortic Valve Disease. Circ Cardiovasc Genet. 2015 Dec;8(6):812-22. doi: 10.1161/CIRCGENETICS.115.001145. Epub 2015 Nov 9. PMID 26553695
- [Background] Dargis N, Lamontagne M, Gaudreault N, Sbarra L, Henry C, Pibarot P, Mathieu P, Bosse Y. Identification of Gender-Specific Genetic Variants in Patients With Bicuspid Aortic Valve. Am J Cardiol. 2016 Feb 1;117(3):420-6. doi: 10.1016/j.amjcard.2015.10.058. Epub 2015 Nov 19. PMID 26708639
- [Background] Mahmut A, Mahjoub H, Boulanger MC, Dahou A, Bouchareb R, Capoulade R, Arsenault BJ, Larose E, Bosse Y, Pibarot P, Mathieu P. Circulating Lp-PLA2 is associated with high valvuloarterial impedance and low arterial compliance in patients with aortic valve bioprostheses. Clin Chim Acta. 2016 Apr 1;455:20-5. doi: 10.1016/j.cca.2016.01.014. Epub 2016 Jan 18. PMID 26797670
- [Background] Capoulade R, Le Ven F, Clavel MA, Dumesnil JG, Dahou A, Thebault C, Arsenault M, O'Connor K, Bedard E, Beaudoin J, Senechal M, Bernier M, Pibarot P. Echocardiographic predictors of outcomes in adults with aortic stenosis. Heart. 2016 Jun 15;102(12):934-42. doi: 10.1136/heartjnl-2015-308742. Epub 2016 Apr 5. PMID 27048774
- [Background] Hadji F, Boulanger MC, Guay SP, Gaudreault N, Amellah S, Mkannez G, Bouchareb R, Marchand JT, Nsaibia MJ, Guauque-Olarte S, Pibarot P, Bouchard L, Bosse Y, Mathieu P. Altered DNA Methylation of Long Noncoding RNA H19 in Calcific Aortic Valve Disease Promotes Mineralization by Silencing NOTCH1. Circulation. 2016 Dec 6;134(23):1848-1862. doi: 10.1161/CIRCULATIONAHA.116.023116. Epub 2016 Oct 27. PMID 27789555
- [Background] Capoulade R, Clavel MA, Le Ven F, Dahou A, Thebault C, Tastet L, Shen M, Arsenault M, Bedard E, Beaudoin J, O'Connor K, Bernier M, Dumesnil JG, Pibarot P. Impact of left ventricular remodelling patterns on outcomes in patients with aortic stenosis. Eur Heart J Cardiovasc Imaging. 2017 Dec 1;18(12):1378-1387. doi: 10.1093/ehjci/jew288. PMID 28064154
- [Background] Tastet L, Enriquez-Sarano M, Capoulade R, Malouf J, Araoz PA, Shen M, Michelena HI, Larose E, Arsenault M, Bedard E, Pibarot P, Clavel MA. Impact of Aortic Valve Calcification and Sex on Hemodynamic Progression and Clinical Outcomes in AS. J Am Coll Cardiol. 2017 Apr 25;69(16):2096-2098. doi: 10.1016/j.jacc.2017.02.037. No abstract available. PMID 28427584
- [Background] Nsaibia MJ, Boulanger MC, Bouchareb R, Mkannez G, Le Quang K, Hadji F, Argaud D, Dahou A, Bosse Y, Koschinsky ML, Pibarot P, Arsenault BJ, Marette A, Mathieu P. OxLDL-derived lysophosphatidic acid promotes the progression of aortic valve stenosis through a LPAR1-RhoA-NF-kappaB pathway. Cardiovasc Res. 2017 Sep 1;113(11):1351-1363. doi: 10.1093/cvr/cvx089. PMID 28472283
- [Background] Shen M, Tastet L, Bergler-Klein J, Pibarot P, Clavel MA. Blood, tissue and imaging biomarkers in calcific aortic valve stenosis: past, present and future. Curr Opin Cardiol. 2018 Mar;33(2):125-133. doi: 10.1097/HCO.0000000000000487. PMID 29194051
- [Background] Theriault S, Gaudreault N, Lamontagne M, Rosa M, Boulanger MC, Messika-Zeitoun D, Clavel MA, Capoulade R, Dagenais F, Pibarot P, Mathieu P, Bosse Y. A transcriptome-wide association study identifies PALMD as a susceptibility gene for calcific aortic valve stenosis. Nat Commun. 2018 Mar 7;9(1):988. doi: 10.1038/s41467-018-03260-6. PMID 29511167
- [Derived] Shen M, Tastet L, Capoulade R, Bedard E, Arsenault M, Clavel MA, Pibarot P. Determinants of Aortic Stenosis Progression in Bicuspid and Tricuspid Aortic Valves. CJC Pediatr Congenit Heart Dis. 2022 Jul 7;1(4):184-192. doi: 10.1016/j.cjcpc.2022.06.004. eCollection 2022 Aug. PMID 37969929
- [Derived] Shen M, Tastet L, Capoulade R, Arsenault M, Bedard E, Clavel MA, Pibarot P. Effect of bicuspid aortic valve phenotype on progression of aortic stenosis. Eur Heart J Cardiovasc Imaging. 2020 Jul 1;21(7):727-734. doi: 10.1093/ehjci/jeaa068. PMID 32386199
- [Derived] Everett RJ, Tastet L, Clavel MA, Chin CWL, Capoulade R, Vassiliou VS, Kwiecinski J, Gomez M, van Beek EJR, White AC, Prasad SK, Larose E, Tuck C, Semple S, Newby DE, Pibarot P, Dweck MR. Progression of Hypertrophy and Myocardial Fibrosis in Aortic Stenosis: A Multicenter Cardiac Magnetic Resonance Study. Circ Cardiovasc Imaging. 2018 Jun;11(6):e007451. doi: 10.1161/CIRCIMAGING.117.007451. PMID 29914867
- [Derived] Pawade T, Clavel MA, Tribouilloy C, Dreyfus J, Mathieu T, Tastet L, Renard C, Gun M, Jenkins WSA, Macron L, Sechrist JW, Lacomis JM, Nguyen V, Galian Gay L, Cuellar Calabria H, Ntalas I, Cartlidge TRG, Prendergast B, Rajani R, Evangelista A, Cavalcante JL, Newby DE, Pibarot P, Messika Zeitoun D, Dweck MR. Computed Tomography Aortic Valve Calcium Scoring in Patients With Aortic Stenosis. Circ Cardiovasc Imaging. 2018 Mar;11(3):e007146. doi: 10.1161/CIRCIMAGING.117.007146. PMID 29555836